CLINICAL TRIAL: NCT06123767
Title: Evaluation of Diagnostic and Predictive Capabilities of Novel Application of Carotid Carotid Stenosis Pressure Gradient Measurement in Patients Undergoing Percutaneous Carotid Angioplasty and Stenting (CAS).
Brief Title: Innovative Application of Pressure Gradient Measurement in Internal Carotid Stenosis in Patients Undergoing CAS
Acronym: NOTICE-CAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Krzysztof Ściborski, Vice-Head of Cath Lab; Department of Cardiology, Center for Heart Disease, 4th Military Hospital, Wrocław, Poland, 4th Military Clinical Hospital with Polyclinic, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ABM/2023/01/00001
Record Dates: First submitted 2023-09-27; First posted 2023-11-09 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Stenting; Stroke
Keywords: CAS (carotid artery stenting); FFR (fractional flow reserve); FFR-CT (Fractional Flow Reserve - Computed Tomography); Carotid Artery Stenosis; Functional assessment of the stenosis; Decision making algorithm
MeSH Terms: conditions — Carotid Stenosis; Stroke; Apraxias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The project is a double-blind study. Neither the researchers nor the participants will know what invasive procedures will be performed on a given patient. Patients, investigators, and all persons involved in performing the procedure or analysis of the data, as well as others with an interest in the study results, will remain blinded to the treatment assigned to individual patients from the beginning of the study until the closure of the database.
  Staff involved in the CAS procedure (with or without blood pressure measurement) will not participate in further patient care and will not provide information to other researchers and people conducting therapy and diagnostics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAS + Intravascular measuring the pressure gradient (Experimental): Patients with internal carotid stenosis qualified for angioplasty with stent implantation.
  Standard CAS procedure with additional intravascular pressure measurements
  Interventions: Procedure: CAS + Intravascular measuring the pressure gradient; Procedure: CAS (standard); Diagnostic Test: Doppler ultrasonound of cephalic arteries; Radiation: Angio-CT of the neck and head; Other: Otolaryngological examination; Other: Psychological examination; Other: Neurological examination; Diagnostic Test: MR cerebral perfusion
- CAS (standard) (Active Comparator): Patients with internal carotid stenosis qualified for angioplasty with stent implantation.
  Standard CAS procedure.
  Interventions: Procedure: CAS (standard); Diagnostic Test: Doppler ultrasonound of cephalic arteries; Radiation: Angio-CT of the neck and head; Other: Otolaryngological examination; Other: Psychological examination; Other: Neurological examination; Diagnostic Test: MR cerebral perfusion

INTERVENTIONS:
Procedure: CAS + Intravascular measuring the pressure gradient — Measurements taken during the procedure during CAS
  * placement of a "FFR"- micro catheter on the neuroprotection wire and taking a measurement before the stenosis and in the internal carotid artery above the stenosis
  * reading the pressure gradient after obtaining a stable value (a minimum of 5 cardiac cycles)
    * the study of intravascular pressure measurements will be performed using a special micro catheter
  Arms: CAS + Intravascular measuring the pressure gradient
Procedure: CAS (standard) — Animation of blood pressure measurements on the "FFR" console without actual measurement in carotid artery ("blinding" of the study to the patient) during CAS procedure.
Diagnostic Test: Doppler ultrasonound of cephalic arteries — non-invasive assessment of carotid stenosis before surgery and assessment of results after CAS (3 and 12 months after CAS)
Radiation: Angio-CT of the neck and head — Non-invasive pre-operative assessment and post-CAS result (3 months after)
Other: Otolaryngological examination — Hearing and balance tests (before and after CAS) - prospective follow-up
Other: Psychological examination — psychological examination with questionnaires (before and after CAS) - prospective follow-up
Other: Neurological examination — neurological examination with questionnaires (before and after CAS) - prospective follow-up
Diagnostic Test: MR cerebral perfusion — Assessment of the cerebral perfusion alterations using DSC (dynamic susceptibility contrast) MR perfusion, before and after CAS (after 3 months):
  Parametric maps of cerebral blood flow (CBF), cerebral blood volume (CBV), time to peak (TTP), and mean transit time (MTT) will be generated and used for the qualitative and quantitative analyses of the following perfusion parameters:
  * cerebral blood volume (CBV) value in ml/100ml;
  * cerebral blood flow (CBF) value in ml/100ml/min;
  * mean transit time (MTT) value in seconds
  * time to peak (TTP) value in seconds

SUMMARY:
About 20% of stroke causes are atherosclerotic strokes caused by carotid artery stenosis.

In 2005, 92% of carotid artery interventions in the USA were performed in asymptomatic patients. It should be noted that screening in the general population for carotid artery disease is unwarranted, due to uncertain eligibility criteria for interventional treatment of asymptomatic patients. On the other hand, 10-15% of all patients with a first-ever stroke will experience an ischemic stroke as a result of previously untreated, asymptomatic, significant carotid artery stenosis.

Carotid artery angioplasty with stent placement (CAS) has become the second method of revascularization. ed, however, there is a great deal of ambiguity in the application of these criteria, which stems from the ratio of the risk to the possible benefit to the patient of performing the procedure, as well as the cost-effectiveness for health care systems.

OBJECTIVES The overall goal is (following the model of measuring fractional flow reserve - FFR) to try to establish a new parameter that could prove helpful in qualifying patients for percutaneous internal carotid artery angioplasty with stent implantation (CAS). Determining whether measuring the pressure gradient across the stenosis will determine which patients will benefit from the CAS procedure. In the absence of convincing evidence on the effects of CAS, especially for so-called asymptomatic patients, it is advisable to establish a parameter that would complement the eligibility criteria that, on the one hand, could prevent strokes in the population of patients with silent internal carotid artery stenosis and, on the other hand, avoid performing the procedure in the absence of benefit.

PRIMARY ENDPOINTS:

1. Assessment of cerebral perfusion by magnetic resonanse before and after CAS
2. Assessment of cognitive symptoms using before and after CAS
3. Assessment of neurological symptoms before and after CAS
4. Assessment of otolaryngological symptoms before and after CAS

SECONDARY ENDPOINTS:

Creation of a non-invasive computed tomography protocol with pressure gradient assessment in patients with carotid artery stenosis.

A final version of the algorithm based on a new diagnostic measurement (concentration gradient) ready to be used in the diagnosis of CAS-eligible patients with an implemented function for automatic classification of measurement results that will indicate the group of patients who will benefit from the CAS procedure.

DETAILED DESCRIPTION:
After qualification for the study (by a neurologist and vascular surgeon), patients meeting properly the inclusion and exclusion criteria will be referred for imaging studies with Doppler ultrasound, angio-CT scan of the arteries of the neck and head and cerebral perfusion in magnetic resonanse (assessment of the cerebral perfusion alterations using DSC (dynamic susceptibility contrast).

In addition, blood will be drawn and stored for subsequent testing. Afterwards, patients qualified for internal carotid artery angioplasty procedures will receive standard saturation treatment with two antiplatelet drugs (acetylsalicylic acid, clopidogrel) before the procedure, strictly according to the guidelines. The procedures are carried out with approved medical equipment (carotid stent, angioplasty balloon, peripheral neuroprotection). The selection of the appropriate equipment used for the procedure depends on the clinical situation, the experience of the operator and the anatomical conditions of the carotid arteries.

Measurements (invasive pressure in carotid artery) taken during the procedure before angioplasty (after insertion of the neuroprotection into the internal carotid artery) and after stent implantation:

COURSE OF THE STUDY

Baseline examination:

* Doppler ultrasound of the extracranial cephalic arteries
* initial qualification for CAS /neurologist, vascular surgeon/
* informed consent to participate in the study
* cardiological consultation (modification of risk factors)
* angio-CT of the neck and head
* assessment of the cerebral perfusion alterations using DSC (dynamic susceptibility contrast) MR perfusion
* additional neurological (with questionnaires), psychological (with questionnaires) and otolaryngological examination
* surgery (CAS) - Department of Vascular Surgery, Department of Cardiology

Measurements (invasive pressure) taken during the procedure before angioplasty (after insertion of the neuroprotection into the internal carotid artery) and after stent implantation:

* placement of a micro catheter to measure invasive pressure
* taking a measurement in the internal carotid artery above the stenosis (in the normal section of this artery)
* performing a measurement before the stenosis (in the normal segment of the common carotid artery at the level of the exit of the external carotid artery)
* reading the pressure gradient after obtaining a stable value (a minimum of 5 cardiac cycles)

  * The study of intravascular pressure measurements will be performed using a special micro catheter of about 1mm in size (i.e., more than 2 times smaller than the delivery system for distal protection, which is the standard procedure, so the risk of complications is minimal). In the study protocol, the insertion of the catheter and measurement of pressures will be followed by the placement of a neuroprotection device in the distal carotid artery (standard of practice) to avoid possible complications.

Evaluation during treatment:

* angio-CT of the neck and head, 3 month after CAS
* assessment of the cerebral perfusion alterations using DSC (dynamic susceptibility contrast) MR perfusion, 3 month after CAS
* Doppler ultrasound of the extracranial cephalic arteries, 3 and 12 month after CAS
* Neurological (with questionnaires), psychological (with questionnaires) and otolaryngological examination betwenn 10-16 week after CAS
* Cardiological evaluation at 3, 6, 12 month after CAS (modification of risk factors)

ELIGIBILITY:
Inclusion Criteria:

* Stenosis of the internal carotid artery in symptomatic patients: > 50%, (confirmed by non-invasive imaging studies: USG, angio-CT), qualified for angioplasty with stent implantation
* Stenosis of the internal carotid artery in asymptomatic patients: >60%, (confirmed by non-invasive imaging studies: USG, angio-CT), qualified for angioplasty with stent implantation
* Age of patients: > 18 years of age
* Provided informed consent to participate in the study.

Exclusion Criteria:

* Inability to obtain informed consent to participate in the study.
* Difficult anatomy of the aortic arch and the descending cephalic arteries (increased atherosclerotic lesions, acute angle of departure of the common carotid arteries, kinking of the internal carotid arteries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Predictive capabilities of the obtained invasive pressure gradient in carotid artery stenosis on changes in cerebral perfusion after surgery | 3 months
  Composite endpoint including:
  Assessment of the predictive capabilities of the obtained pressure gradient values
  * on changes in cerebral perfusion after surgery (assessment of the cerebral perfusion alterations using DSC (dynamic susceptibility contrast) MR perfusion, before and after CAS
Predictive capabilities of the obtained invasive pressure gradient in carotid artery stenosis on neurological status | 12 months
  Composite endpoint including:
  - changes in neurological status (assesed by the MMSE, mini-mental state examination; NIHSS, National Institutes of Health Stroke Scale),
Predictive capabilities of the obtained invasive pressure gradient in carotid artery stenosis on mental status | 12 months
  Composite endpoint including:
  - changes in cognitive functions (assesed by the MOCA, Montreal Cognitive Assessment - test)
Predictive capabilities of the obtained invasive pressure gradient in carotid artery stenosis on otolaryngological status in hearing functions | 12 months
  Composite endpoint including:
  - changes in hearing functions (assesed by the audiometry, tympanometry and ipsilateral middle ear reflex, otoemission, Skarzynski Tinnitus Scale, ABR - Auditory Brainstem Response, BERA)
Predictive capabilities of the obtained invasive pressure gradient in carotid artery stenosis on otolaryngological status in labyrinth functions | 12 months
  Composite endpoint including:
  - changes in labyrinth functions (assesed by the Skarzynski Tinnitus Scale)
Predictive capabilities of the obtained invasive pressure gradient in carotid artery stenosis on MACEs after surgery | 12 months
  Composite endpoint including:
  - occurence of stroke/TIA or death
Repeatability the diagnostic possibilities of non-invasive tests (Doppler ultrasound) in invasive pressure gradient values | 12 months
  Composite endpoint including:
  - comparison of the obtained invasive pressure gradient values with Doppler ultrasound (PSV, peak systolic velocity; EDV, end-diastolic velocity; estimated degree of stenosis)
Repeatability the diagnostic possibilities of non-invasive tests (CT angiogram) in invasive pressure gradient values | 12 months
  Composite endpoint including:
  - comparison of the obtained invasive pressure gradient values with angio-CT: degree of stenosis
Repeatability the diagnostic possibilities of non-invasive tests ("CT-FFR") in invasive pressure gradient values | 12 months
  Composite endpoint including:
  - comparison of the obtained invasive pressure gradient values with "CT-FFR" (planned creation of an algorithm based on test results: invasive pressure gradient, Doppler ultrasound, angio-CT)
Incidence of Treatment-Related Adverse Events [safety and tolerability] associated with the invasive intravascular pressure measurement procedure (1) | 12 months
  Composite endpoint including:
  - occurrence of periprocedural neurological event: TIA, stroke, death in patients who underwent CAS with the invasive intravascular pressure measurement procedure
Incidence of Treatment-Related Adverse Events [safety and tolerability] associated with the invasive intravascular pressure measurement procedure (2) | 12 months
  Composite endpoint including:
  - occurrence of another periprocedural complication: vascular spasm, perforation, cardiac arrhythmia, hypotonia/hypertension in patients who underwent CAS with the invasive intravascular pressure measurement procedure
Incidence of Treatment-Related Adverse Events [safety and tolerability] associated with the invasive intravascular pressure measurement procedure (3) | 12 months
  Composite endpoint including:
  - occurrence of new hypodense (impact) foci in the head CT scan after the procedure in patients who underwent CAS with the invasive intravascular pressure measurement procedure
Incidence of Treatment-Related Adverse Events [safety and tolerability] associated with the invasive intravascular pressure measurement procedure (4) | 12 months
  Composite endpoint including:
  - changes (improvement or deterioration) in brain perfusion (see point 1.) in the post-operative examination in patients who underwent CAS with the invasive intravascular pressure measurement procedure

SECONDARY OUTCOMES:
Algorithm angio-CT/non invasive pressure measurement in carotid | 48 months
  Creation a multiple regression model based on the data from non-invasive pre-procedural measurements on the incidence of unfavourable outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Ściborski, MD, PhD, Principal Investigator — 4th Military Hospital in Wrocław; Waldemar Banasiak, MD, PhD, Study Director — 4th Military Hospital in Wrocław; Artur Telichowski, MD, PhD, Study Director — 4th Military Clinical Hospital with Polyclinic, Poland; Adrian Doroszko, MD, PhD, Study Director — 4th Military Clinical Hospital with Polyclinic, Poland
Locations (1):
- 4th Military Hospital, Wroclaw, Lower Silesian Voivodeship, Poland

REFERENCES:
- [Background] Patel MR, Calhoon JH, Dehmer GJ, Grantham JA, Maddox TM, Maron DJ, Smith PK. ACC/AATS/AHA/ASE/ASNC/SCAI/SCCT/STS 2017 Appropriate Use Criteria for Coronary Revascularization in Patients With Stable Ischemic Heart Disease: A Report of the American College of Cardiology Appropriate Use Criteria Task Force, American Association for Thoracic Surgery, American Heart Association, American Society of Echocardiography, American Society of Nuclear Cardiology, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Computed Tomography, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2017 May 2;69(17):2212-2241. doi: 10.1016/j.jacc.2017.02.001. Epub 2017 Mar 10. No abstract available. PMID 28291663
- [Background] Christou MA, Siontis GC, Katritsis DG, Ioannidis JP. Meta-analysis of fractional flow reserve versus quantitative coronary angiography and noninvasive imaging for evaluation of myocardial ischemia. Am J Cardiol. 2007 Feb 15;99(4):450-6. doi: 10.1016/j.amjcard.2006.09.092. Epub 2006 Dec 20. PMID 17293182
- [Background] Curzen N, Rana O, Nicholas Z, Golledge P, Zaman A, Oldroyd K, Hanratty C, Banning A, Wheatcroft S, Hobson A, Chitkara K, Hildick-Smith D, McKenzie D, Calver A, Dimitrov BD, Corbett S. Does routine pressure wire assessment influence management strategy at coronary angiography for diagnosis of chest pain?: the RIPCORD study. Circ Cardiovasc Interv. 2014 Apr;7(2):248-55. doi: 10.1161/CIRCINTERVENTIONS.113.000978. Epub 2014 Mar 18. PMID 24642999
- [Background] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO. [2018 ESC/EACTS Guidelines on myocardial revascularization]. Kardiol Pol. 2018;76(12):1585-1664. doi: 10.5603/KP.2018.0228. No abstract available. Polish. PMID 30566213
- [Background] Van't Veer M, Pijls NHJ, Hennigan B, Watkins S, Ali ZA, De Bruyne B, Zimmermann FM, van Nunen LX, Barbato E, Berry C, Oldroyd KG. Comparison of Different Diastolic Resting Indexes to iFR: Are They All Equal? J Am Coll Cardiol. 2017 Dec 26;70(25):3088-3096. doi: 10.1016/j.jacc.2017.10.066. PMID 29268922
- [Background] Svanerud J, Ahn JM, Jeremias A, van 't Veer M, Gore A, Maehara A, Crowley A, Pijls NHJ, De Bruyne B, Johnson NP, Hennigan B, Watkins S, Berry C, Oldroyd KG, Park SJ, Ali ZA. Validation of a novel non-hyperaemic index of coronary artery stenosis severity: the Resting Full-cycle Ratio (VALIDATE RFR) study. EuroIntervention. 2018 Sep 20;14(7):806-814. doi: 10.4244/EIJ-D-18-00342. PMID 29790478
- [Background] Taylor CA, Fonte TA, Min JK. Computational fluid dynamics applied to cardiac computed tomography for noninvasive quantification of fractional flow reserve: scientific basis. J Am Coll Cardiol. 2013 Jun 4;61(22):2233-41. doi: 10.1016/j.jacc.2012.11.083. Epub 2013 Apr 3. PMID 23562923
- [Background] Min JK, Taylor CA, Achenbach S, Koo BK, Leipsic J, Norgaard BL, Pijls NJ, De Bruyne B. Noninvasive Fractional Flow Reserve Derived From Coronary CT Angiography: Clinical Data and Scientific Principles. JACC Cardiovasc Imaging. 2015 Oct;8(10):1209-1222. doi: 10.1016/j.jcmg.2015.08.006. PMID 26481846
- [Background] Rothwell PM, Eliasziw M, Gutnikov SA, Fox AJ, Taylor DW, Mayberg MR, Warlow CP, Barnett HJ; Carotid Endarterectomy Trialists' Collaboration. Analysis of pooled data from the randomised controlled trials of endarterectomy for symptomatic carotid stenosis. Lancet. 2003 Jan 11;361(9352):107-16. doi: 10.1016/s0140-6736(03)12228-3. PMID 12531577
- [Background] Mas JL, Chatellier G, Beyssen B, Branchereau A, Moulin T, Becquemin JP, Larrue V, Lievre M, Leys D, Bonneville JF, Watelet J, Pruvo JP, Albucher JF, Viguier A, Piquet P, Garnier P, Viader F, Touze E, Giroud M, Hosseini H, Pillet JC, Favrole P, Neau JP, Ducrocq X; EVA-3S Investigators. Endarterectomy versus stenting in patients with symptomatic severe carotid stenosis. N Engl J Med. 2006 Oct 19;355(16):1660-71. doi: 10.1056/NEJMoa061752. PMID 17050890
- [Background] SPACE Collaborative Group; Ringleb PA, Allenberg J, Bruckmann H, Eckstein HH, Fraedrich G, Hartmann M, Hennerici M, Jansen O, Klein G, Kunze A, Marx P, Niederkorn K, Schmiedt W, Solymosi L, Stingele R, Zeumer H, Hacke W. 30 day results from the SPACE trial of stent-protected angioplasty versus carotid endarterectomy in symptomatic patients: a randomised non-inferiority trial. Lancet. 2006 Oct 7;368(9543):1239-47. doi: 10.1016/S0140-6736(06)69122-8. PMID 17027729
- [Background] International Carotid Stenting Study investigators; Ederle J, Dobson J, Featherstone RL, Bonati LH, van der Worp HB, de Borst GJ, Lo TH, Gaines P, Dorman PJ, Macdonald S, Lyrer PA, Hendriks JM, McCollum C, Nederkoorn PJ, Brown MM. Carotid artery stenting compared with endarterectomy in patients with symptomatic carotid stenosis (International Carotid Stenting Study): an interim analysis of a randomised controlled trial. Lancet. 2010 Mar 20;375(9719):985-97. doi: 10.1016/S0140-6736(10)60239-5. Epub 2010 Feb 25. PMID 20189239
- [Background] Brott TG, Hobson RW 2nd, Howard G, Roubin GS, Clark WM, Brooks W, Mackey A, Hill MD, Leimgruber PP, Sheffet AJ, Howard VJ, Moore WS, Voeks JH, Hopkins LN, Cutlip DE, Cohen DJ, Popma JJ, Ferguson RD, Cohen SN, Blackshear JL, Silver FL, Mohr JP, Lal BK, Meschia JF; CREST Investigators. Stenting versus endarterectomy for treatment of carotid-artery stenosis. N Engl J Med. 2010 Jul 1;363(1):11-23. doi: 10.1056/NEJMoa0912321. Epub 2010 May 26. PMID 20505173
- [Background] Bonati LH, Jongen LM, Haller S, Flach HZ, Dobson J, Nederkoorn PJ, Macdonald S, Gaines PA, Waaijer A, Stierli P, Jager HR, Lyrer PA, Kappelle LJ, Wetzel SG, van der Lugt A, Mali WP, Brown MM, van der Worp HB, Engelter ST; ICSS-MRI study group. New ischaemic brain lesions on MRI after stenting or endarterectomy for symptomatic carotid stenosis: a substudy of the International Carotid Stenting Study (ICSS). Lancet Neurol. 2010 Apr;9(4):353-62. doi: 10.1016/S1474-4422(10)70057-0. Epub 2010 Feb 25. PMID 20189458
- [Background] Schnaudigel S, Groschel K, Pilgram SM, Kastrup A. New brain lesions after carotid stenting versus carotid endarterectomy: a systematic review of the literature. Stroke. 2008 Jun;39(6):1911-9. doi: 10.1161/STROKEAHA.107.500603. Epub 2008 Apr 3. PMID 18388346
- [Background] McPhee JT, Schanzer A, Messina LM, Eslami MH. Carotid artery stenting has increased rates of postprocedure stroke, death, and resource utilization than does carotid endarterectomy in the United States, 2005. J Vasc Surg. 2008 Dec;48(6):1442-50, 1450.e1. doi: 10.1016/j.jvs.2008.07.017. Epub 2008 Oct 1. PMID 18829236
- [Background] Naylor AR. Why is the management of asymptomatic carotid disease so controversial? Surgeon. 2015 Feb;13(1):34-43. doi: 10.1016/j.surge.2014.08.004. Epub 2014 Oct 14. PMID 25439170
- [Background] Hadar N, Raman G, Moorthy D, O'Donnell TF, Thaler DE, Feldmann E, Lau J, Kitsios GD, Dahabreh IJ. Asymptomatic carotid artery stenosis treated with medical therapy alone: temporal trends and implications for risk assessment and the design of future studies. Cerebrovasc Dis. 2014;38(3):163-73. doi: 10.1159/000365206. Epub 2014 Oct 9. PMID 25300534
- [Background] Endarterectomy for asymptomatic carotid artery stenosis. Executive Committee for the Asymptomatic Carotid Atherosclerosis Study. JAMA. 1995 May 10;273(18):1421-8. PMID 7723155
- [Background] Baker WH, Howard VJ, Howard G, Toole JF. Effect of contralateral occlusion on long-term efficacy of endarterectomy in the asymptomatic carotid atherosclerosis study (ACAS). ACAS Investigators. Stroke. 2000 Oct;31(10):2330-4. doi: 10.1161/01.str.31.10.2330. PMID 11022059